CLINICAL TRIAL: NCT06166381
Title: Parenteral Versus Combined Parenteral With Vancomycin-soaked Graft in Decreasing the Risk of Infection in ACL Reconstruction Surgery: A Randomized Controlled Trial
Brief Title: Parenteral Versus Combined Parenteral With Vancomycin-soaked Graft in ACL Reconstruction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Duhok (Other)
Responsible Party: Principal Investigator, Jagar Omar Doski, Assistant Professor, University of Duhok
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 123456789
Record Dates: First submitted 2023-12-04; First posted 2023-12-12 (Actual); Last update posted 2024-12-30 (Actual); Status verified 2024-12

CONDITIONS: Infection, Bacterial
Keywords: Anterior cruciate ligament; reconstruction; infection; vancomycin presoaked graft
MeSH Terms: conditions — Bacterial Infections; Infections | interventions — Ceftriaxone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): This group will receive parenteral antibiotics to prevent infection in the surgery.
  Interventions: Drug: Parenteral Antibacterial Agents
- clinical trial (Experimental): This group will include patients who will receive parenteral antibiotics combined with vancomycin presoaked solution for the graft.
  Interventions: Drug: Parenteral Antibacterial Agents; Drug: Parenteral Antibacterial Agents plus Vancomycin pre-soaked graft

INTERVENTIONS:
Drug: Parenteral Antibacterial Agents — Parenteral antibiotic (ceftriaxone) 1 g to be given in 3 doses, at induction of anesthesia, 12 hours postoperative, and 24 hours postoperative.
  Other Names: Ceftriaxone sodium
Drug: Parenteral Antibacterial Agents plus Vancomycin pre-soaked graft — in addition to the parenteral ceftriaxone intravenous injections, the ACL graft will be soaked in the vancomycin solution for 20 minutes when prepared outside the body of patient.
  Other Names: Ceftriaxone sodium intravenously plus Vancomycin pre-soaked graft
  Arms: clinical trial

SUMMARY:
An anterior cruciate ligament (ACL) tear is one of the knee joint's most common soft tissue injuries [1]. It is frequently injured in non-contact and some contact competition sports and even during ordinary life activities. With an annual incidence of 68.6 per 100,000 person-years, ACL tears remain a common orthopedic injury [2]. Females are two to eight times more likely to develop ACL tears in sports compared to men who play the same particular sports [3]. Most highly demanding persons and those who develop frequent instability of their knee require reconstructive surgery on the ACL to prevent early degenerative changes in their knees. This is done by completely removing the torn or ruptured ACL and replacement with a piece of tendon or ligament (graft) [4].

Post-operative infection may occur in 0.14-2.6% of ACL reconstruction despite intravenous antibiotics prophylaxis [5,6]. The deep infection results in poor outcomes with pain, stiffness, arthrofibrosis, and articular cartilage degeneration [7,8]. Few studies reported improved outcomes of infection control when the autograft presoaked in vancomycin solution during the preparation process outside the body before being transferred to the knee of the patient [9-13]. Systematic reviews and meta-analysis showed that all the articles discussing the outcome of vancomycin presoaked autograft in ACL reconstruction surgery were case series, observational retrospective, prospective comparative, or case-control studies [14,15]. Randomized control trial (RCT) provides the strongest evidence among the primary research studies to confirm the effectiveness of a new method of treatment [16,17]. To date, there is no available RCT study in this field.

DETAILED DESCRIPTION:
Aim This study aims to do RTC research on the role of vancomycin-presoaked autograft in ACL reconstruction to decrease the risk of infection.

Objectives To treat patients undergoing ACL reconstruction surgery by two methods to prevent infection (parenteral antibiotic and combined parenteral antibiotic with vancomycin presoaked autograft). To compare between odds ratio of infection occurrence. To check the superiority of the added vancomycin presoaked method in decreasing the risk of infection.

Methods Study type It will be a randomized controlled clinical trial of superiority type. It will be based on a parallel-group type with an allocation ratio of 1:1.

Study setting The research will be conducted in the orthopedic unit, at Azadi Teaching Hospital, Duhok, Iraq.

Inclusion criteria Patients between the ages of 20 to 45 years, of any sex, with ACL dysfunction and needing ACL reconstruction surgery, will be involved in this research.

Exclusion criteria Patients for revision surgery of ACL reconstruction, inflammatory rheumatological disorders, and refusal to participate in the study.

Interventions The patients will be divided into 2 groups: group one (control) will be those who will receive only parenteral antibiotics at induction of anesthesia and for 5 days after the operation. The second group (trial) will receive parenteral antibiotics combined with soaking the autograft of ACL autograft into the vancomycin solution duration preparation of the graft recipient site.

Outcomes The primary outcome will be the odds of cases developing signs of infection up to 6 months postoperatively. No secondary outcome will be recorded for this study.

Sample size The assumed sample size was calculated by using the G*Power 3.1.9.7 computer software program. A minimum of 288 participants (144 for each group) are required to have an 80% chance of detecting the difference between the groups with a two-sided 95% confidence level (0.05 level of significance) to achieve a difference in the odds ratio of 1.8.

Randomization

The allocation of the participants into the modalities of the treatment will be done by a simple randomization method with an allocation ratio of 1:1. It will be generated by using the website program www.randomization.com.

Statistical analysis The data analysis will be performed by SPSS 23.0. The statistical analysis will include the standard descriptive statistics used to describe the basic descriptive data of the patients. The means and standard deviations (SD) or medians and interquartile ranges were used for the continuous variables, while frequencies and percentages were used for the categorical variables. The comparison between the outcomes of the treatment modalities in both groups will be done by finding the difference between the summary statistics in the Chi-squared test. The difference will be considered statistically significant when the p-value is less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

* ACL injury that interferes with life activities and/or sports

Exclusion Criteria:

* Patients for revision surgery of ACL reconstruction
* patients with inflammatory rheumatological disorders
* Refusal to participate in the study.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Estimated)
Dates: Start 2024-01-25 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
infection | 1st day postoperative upto 6 months
  deep infection occurs around the graft of the ACL

CONTACTS AND LOCATIONS:
Locations (1):
- College of Medicine/University of Duhok, Duhok, Iraq

IPD SHARING:
Plan to Share IPD: Yes
The information will be supplied to other researches on reasonable request.
Supporting Information: Study Protocol, SAP
Time Frame: from the time of publication of the article and up to 5 years after.
Access Criteria: email request

REFERENCES:
- [Result] Cimino F, Volk BS, Setter D. Anterior cruciate ligament injury: diagnosis, management, and prevention. Am Fam Physician. 2010 Oct 15;82(8):917-22. PMID 20949884
- [Result] Sanders TL, Maradit Kremers H, Bryan AJ, Larson DR, Dahm DL, Levy BA, Stuart MJ, Krych AJ. Incidence of Anterior Cruciate Ligament Tears and Reconstruction: A 21-Year Population-Based Study. Am J Sports Med. 2016 Jun;44(6):1502-7. doi: 10.1177/0363546516629944. Epub 2016 Feb 26. PMID 26920430
- [Result] Faryniarz DA, Bhargava M, Lajam C, Attia ET, Hannafin JA. Quantitation of estrogen receptors and relaxin binding in human anterior cruciate ligament fibroblasts. In Vitro Cell Dev Biol Anim. 2006 Jul-Aug;42(7):176-81. doi: 10.1290/0512089.1. PMID 16948498
- [Result] Bansal A, Lamplot JD, VandenBerg J, Brophy RH. Meta-analysis of the Risk of Infections After Anterior Cruciate Ligament Reconstruction by Graft Type. Am J Sports Med. 2018 May;46(6):1500-1508. doi: 10.1177/0363546517714450. Epub 2017 Jul 24. PMID 28737955
- [Result] Maletis GB, Inacio MC, Reynolds S, Desmond JL, Maletis MM, Funahashi TT. Incidence of postoperative anterior cruciate ligament reconstruction infections: graft choice makes a difference. Am J Sports Med. 2013 Aug;41(8):1780-5. doi: 10.1177/0363546513490665. Epub 2013 Jun 7. PMID 23749343
- [Result] Schub DL, Schmitz LM, Sakamoto FA, Winalski CS, Parker RD. Long-term outcomes of postoperative septic arthritis after anterior cruciate ligament reconstruction. Am J Sports Med. 2012 Dec;40(12):2764-70. doi: 10.1177/0363546512461903. Epub 2012 Oct 19. PMID 23087081
- [Result] Stucken C, Garras DN, Shaner JL, Cohen SB. Infections in anterior cruciate ligament reconstruction. Sports Health. 2013 Nov;5(6):553-7. doi: 10.1177/1941738113489099. PMID 24427432
- [Result] Vertullo CJ, Quick M, Jones A, Grayson JE. A surgical technique using presoaked vancomycin hamstring grafts to decrease the risk of infection after anterior cruciate ligament reconstruction. Arthroscopy. 2012 Mar;28(3):337-42. doi: 10.1016/j.arthro.2011.08.301. Epub 2011 Nov 23. PMID 22112612
- [Result] Perez-Prieto D, Torres-Claramunt R, Gelber PE, Shehata TMA, Pelfort X, Monllau JC. Autograft soaking in vancomycin reduces the risk of infection after anterior cruciate ligament reconstruction. Knee Surg Sports Traumatol Arthrosc. 2016 Sep;24(9):2724-2728. doi: 10.1007/s00167-014-3438-y. Epub 2014 Nov 22. PMID 25416672
- [Result] Phegan M, Grayson JE, Vertullo CJ. No infections in 1300 anterior cruciate ligament reconstructions with vancomycin pre-soaking of hamstring grafts. Knee Surg Sports Traumatol Arthrosc. 2016 Sep;24(9):2729-2735. doi: 10.1007/s00167-015-3558-z. Epub 2015 Mar 14. PMID 25771788
- [Result] Carrozzo A, Saithna A, Ferreira A, Guy S, Chadli L, Monaco E, Perez-Prieto D, Bohu Y, Vieira TD, Sonnery-Cottet B. Presoaking ACL Grafts in Vancomycin Decreases the Frequency of Postoperative Septic Arthritis: A Cohort Study of 29,659 Patients, Systematic Review, and Meta-analysis From the SANTI Study Group. Orthop J Sports Med. 2022 Feb 7;10(2):23259671211073928. doi: 10.1177/23259671211073928. eCollection 2022 Feb. PMID 35155711
- [Result] Bohu Y, Klouche S, Sezer HB, Herman S, Grimaud O, Gerometta A, Meyer A, Lefevre N. Vancomycin-soaked autografts during ACL reconstruction reduce the risk of post-operative infection without affecting return to sport or knee function. Knee Surg Sports Traumatol Arthrosc. 2020 Aug;28(8):2578-2585. doi: 10.1007/s00167-020-05879-9. Epub 2020 Feb 5. PMID 32025764
- [Result] Hu M, Zhang Y, Shang G, Guo J, Xu H, Ma X, Yang X, Xiang S. Vancomycin presoak reduces infection in anterior cruciate ligament reconstruction: a systematic review and meta-analysis. BMC Musculoskelet Disord. 2023 Apr 5;24(1):267. doi: 10.1186/s12891-023-06331-y. PMID 37020216
- [Result] Rodriguez-Merchan EC, Ribbans WJ. The role of vancomycin-soaking of the graft in anterior cruciate ligament reconstruction. J ISAKOS. 2022 Apr;7(2):94-98. doi: 10.1016/j.jisako.2021.12.006. Epub 2022 Jan 7. PMID 35546439
- [Result] Murad MH, Asi N, Alsawas M, Alahdab F. New evidence pyramid. Evid Based Med. 2016 Aug;21(4):125-7. doi: 10.1136/ebmed-2016-110401. Epub 2016 Jun 23. PMID 27339128
- [Result] Kapoor MC. Types of studies and research design. Indian J Anaesth. 2016 Sep;60(9):626-630. doi: 10.4103/0019-5049.190616. PMID 27729687